CLINICAL TRIAL: NCT07111884
Title: National, Observational, Non-interventional, Retro- and Prospective Clinical Multiple Myeloma Registry GMMG
Brief Title: GMMG Multiple Myeloma Registry
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Hartmut Goldschmidt (Other)
Collaborators: Dietmar Hopp Stiftung (Other); KKS Netzwerk (Network); German Cancer Research Center (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Hartmut Goldschmidt, Head of GMMG- study group, University of Heidelberg Medical Center
Organization: University of Heidelberg Medical Center (Other)
Other Study IDs: GMMG Myeloma Registry; DRKS00026970 (Registry Identifier: German Clinical Trials Registry)
Record Dates: First submitted 2024-07-30; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: registry; longtime follow-up; elotuzumab; real world data
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with multiple myeloma: newly- diagnosed, transplant eligible multiple myeloma patients

SUMMARY:
The goal of this observational study is to collect long-term clinical follow-up data on patients with multiple myeloma who participated in a therapy study of the German-Speaking Myeloma Multicenter Group (GMMG). Target variables of interest are:

Overall survival, progression-free survival and follow-up time.

The relevant registry data will be provided and evaluated together with the therapy study data for scientific research projects.

This allows seamless documentation of patient data from the end of the trial to long-term follow-up.

DETAILED DESCRIPTION:
The German-speaking Myeloma Multicenter Group (GMMG) registry is a national, observational, non-interventional, retro-and prospective clinical myeloma registry of multiple myeloma patients in Germany. The registry includes the study database of the prospective trials led by the GMMG, with basic data, diagnosis, therapy and longtime follow-up. The sample size is unlimited.

The Myeloma Registry was activated on December 8, 2022. Currently 35 GMMG centers in Germany are participating. The first longtime follow-up data set included in the registry was the GMMG-HD 6 trial. The GMMG-HD6 trial is a phase 3 trial which investigated the efficacy of the addition of the anti-SLAMF7 monoclonal antibody, elotuzumab, to the standard induction and consolidation therapy consisting of lenalidomide, bortezomib and dexamethasone in transplant-eligible patients with newly diagnosed multiple myeloma.

Target variables of interest are progression-free survival (PFS) from randomization, overall survival (OS), the follow-up time, the cause of death and the therapy free time after first relapse and its treatment. Further objectives will be defined and analyzed for each evaluation.

Participations will be observed while the patient is being treated with standard of care until death, lost to follow-up or consent withdrawn. Follow-ups will be documented every six months until the 1st Progression Disease and then annually. The pseudonymized clinical data is stored in a separate database (eCRF) and is monitored centrally on a regular basis. The eCRF contain automated plausibility checks, so called queries.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in a a therapy study of the GMMG study group

Exclusion Criteria:

* patients with organ amyloidosis at time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly-diagnosed, transplant-eligible multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
progression free survival | after 5 years, and then through study completion, an average of 1 year

OTHER OUTCOMES:
overall survival | after 5 years, and then through study completion, an average of 1 year
follow-up time | after 5 years, and then through study completion, an average of 1 year
  The follow-up time of a patient in the ITT is estimated using the reverse Kaplan-Meier method. It is defined as the time from the date of randomization to the last known contact.
cause of death | after 5 years, and then through study completion, an average of 1 year
therapy free time after first relapse and its treatment | after 5 years, and then through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, Prof., Principal Investigator — University Hospital Heidelberg
Locations (35):
- Germany (35):
  - HELIOS Klinikum, Klinik für Hämatologie, Onkologie und Immunologie, Berlin
  - Charité Campus Benjamin Franklin, III. Med. Abt. (Hämatologie/Onkologie), Berlin
  - Klinikum Bielefeld, Klinik für Hämatologie, Onkologie und Palliativmedizin, Bielefeld
  - Medizinische Universitätsklinik, Knappschaftskrankenhaus, Bochum
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik III, Schwerpunkt Onkologie, Hämatologie und Rheumatologie, Bonn
  - Klinikum Chemnitz GmbH, Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln, Klinik I - Innere Medizin, Cologne
  - Onkologisches Studienzentrum Darmstadt, Darmstadt
  - Klinikum Darmstadt, Med. Klinik V, Hämatologie/Onkologie, Darmstadt
  - Universitätsklinikum Düsseldorf, Klinik für Hämatologie,Onkologie und Klin. Immunologie, Düsseldorf
  - Universitätsklinik Erlangen, Erlangen
  - Universitätsklinikum Essen, Klinik für Hämatologie und Stammzelltransplantation, Essen
  - Ev. Krankenhaus Essen-Werden gGmbH, Zentrum für Innere Medizin, Klinik für Hämatologie, Onkologie und Stammzelltransplantation, Essen
  - Universitätsklinikum Frankfurt, Goethe-Universität Medizinische Klinik II, Frankfurt am Main
  - Justus-Liebig-Universität, Medizinische Klinik IV, Giessen
  - Kath. Krankenhaus Hagen GmbH, Abt. Hämatologie/Onkologie, Hagen
  - Asklepios Klinik Hamburg Altona, II. Med. Klinik, Hamburg
  - Onkologische Schwerpunktpraxis, Heidelberg
  - University Hospital Heidelberg, Med. Klinik V, Heidelberg
  - SLK Kliniken Heilbronn, Med. Klinik III, Heilbronn
  - Universitätsklinikum des Saarlandes, Innere Medizin I, Homburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Praxisklinik für Hämatologie und Onkologie, Koblenz
  - Onkologisches Zentrum, Gemeinschaftspraxis f. Hämatologie u. Onkologie im Caritas KH, Lebach
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, III. Med. Klinik, Mainz
  - III. Medizinische Klinik Hämatologie und Internistische Onkologie, Mannheim
  - Mannheimer Onkologie Praxis, Mannheim
  - Philipps-Universität Marburg, Hämatologie/Onkologie/Immunologie, Marburg
  - Krankenhaus Maria Hilf GmbH, Franziskuskrankenhaus, Med. Klinik I, Mönchengladbach
  - Krankenhaus Barmherzige Brüder, Klinik für Onkologie und Hämatologie, Regensburg
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Innere Medizin III, Schwäbisch Hall
  - ZAHO-Zentrum für ambulante Hämatologie und Onkologie, Standort Siegburg, Siegburg
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - University Hospital Tübingen, Med. Klinik und Poliklinik, Abt. II, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
Publications
Supporting Information: Study Protocol, ICF
Time Frame: anticipated after end registry